CLINICAL TRIAL: NCT05382182
Title: Outcome Of Treatment Of Prostate Cancer at Sohag University Hospital Between 2017 to 2021
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Sayed, resident doctor at oncology department at faculty of medicine sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-05-03
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: androgen deprivation therapy — outcome of hormonal treatment as androgen deprivation therapy on prostate cancer patient on survival and relapse
Radiation: external beam radiotherapy — outcome of radiotherapy as external beam radiotherapy on prostate cancer patient on survival and relapse

SUMMARY:
Worldwide, prostate cancer is the most commonly diagnosed male cancer and the fourth leading cause of cancer death in men. Risk stratification is according to cancer stage, Gleason score, and PSA level .

Definitive treatment of localized disease ( low and favorable intermediate risk) includes watchful waiting , active surveillance , radiation therapy , radical prostatectomy and cryotherapy .Primary treatment of unfavorable intermediate risk , high risk localized disease and locally advanced prostate cancer , includes both radical prostatectomy (RP) and EBRT + long-term androgen deprivation therapy (ADT) .Treatment options of metastatic prostate cancer include pain medications, bisphosphonates, hormonal treatment, chemotherapy, radiotherapy, immunotherapy, focused radiation, and other targeted therapies .

ELIGIBILITY:
Inclusion Criteria:

* Patients at age of 18 years old and above.
* All stages and grades of prostate cancer.
* Epithelial types of prostate cancer.

Exclusion Criteria:

* Age below 18 years old.
* Presence of other malignancies.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: prostate cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 6 months
  Overall survival defined as the time from the date of diagnosis to the last date seen .
progression free survival | 6 months
  Progression-free survival defined as the length of time during and after the treatment of cancer that a patient lives with the disease but it does not get worse.
disease free survival | 6 months
  Disease free survival defined as the time from the end of treatment to the date of first relapse .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Costello LC, Franklin RB. A comprehensive review of the role of zinc in normal prostate function and metabolism; and its implications in prostate cancer. Arch Biochem Biophys. 2016 Dec 1;611:100-112. doi: 10.1016/j.abb.2016.04.014. Epub 2016 Apr 27. PMID 27132038
- [Background] Herden J, Heidenreich A, Weissbach L. [TNM-Classification of localized prostate cancer : The clinical T-category does not correspond to the required demands]. Urologe A. 2016 Dec;55(12):1564-1572. doi: 10.1007/s00120-016-0264-5. German. PMID 27830286
- [Background] Moris L, Cumberbatch MG, Van den Broeck T, Gandaglia G, Fossati N, Kelly B, Pal R, Briers E, Cornford P, De Santis M, Fanti S, Gillessen S, Grummet JP, Henry AM, Lam TBL, Lardas M, Liew M, Mason MD, Omar MI, Rouviere O, Schoots IG, Tilki D, van den Bergh RCN, van Der Kwast TH, van Der Poel HG, Willemse PM, Yuan CY, Konety B, Dorff T, Jain S, Mottet N, Wiegel T. Benefits and Risks of Primary Treatments for High-risk Localized and Locally Advanced Prostate Cancer: An International Multidisciplinary Systematic Review. Eur Urol. 2020 May;77(5):614-627. doi: 10.1016/j.eururo.2020.01.033. Epub 2020 Mar 4. PMID 32146018
- [Background] Verma S, Choyke PL, Eberhardt SC, Oto A, Tempany CM, Turkbey B, Rosenkrantz AB. The Current State of MR Imaging-targeted Biopsy Techniques for Detection of Prostate Cancer. Radiology. 2017 Nov;285(2):343-356. doi: 10.1148/radiol.2017161684. PMID 29045233